CLINICAL TRIAL: NCT05964855
Title: Comparison of Various Prosthetic Foot-Ankle Mechanisms
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2306001029
Record Dates: First submitted 2023-07-11; First posted 2023-07-28 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Transtibial Amputation - Unilateral
Keywords: Foot-ankle device; prosthesis; mobility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Unilateral Subject Group (Experimental): Foot-ankle devices will be given to this group to evaluate and compare the devices.
  Interventions: Device: MIT Variable Stiffness Prosthesis; Device: MIT Variable Equilibrium Angle Prosthesis; Device: MIT Sliding Beam Passive Prosthesis; Device: Ossur Pro-flex XC; Device: Blatchford Elan Variable-Dampening Prosthesis

INTERVENTIONS:
Device: MIT Variable Stiffness Prosthesis — Proprietary electronically-controlled prosthesis that can vary its effective stiffness.
Device: MIT Variable Equilibrium Angle Prosthesis — Proprietary manually-controlled prosthesis that can vary its effective ankle equilibrium angle.
Device: MIT Sliding Beam Passive Prosthesis — Proprietary fixed-stiffness passive foot-ankle prosthesis.
Device: Ossur Pro-flex XC — Commercially-available passive fixed-stiffness foot-ankle prosthesis by Ossur.
Device: Blatchford Elan Variable-Dampening Prosthesis — Commercially-available electronically-controlled prosthesis that can vary its effective dampening.
  Other Names: Elan

SUMMARY:
In summary, subjects will be asked to wear a number of sensors and use different ankle-foot prostheses in place of their customary prosthesis. Data will be collected from the wearable sensors, VICON motion capture system, video cameras, and force sensors in the ground as they walk on level-ground, on a treadmill, and on stairs. The controller of any powered prosthesis will be electronically adjusted between trials or while the subject walks to determine how their gait changes in response to these changes. Trials will also be conducted with a standard passive prosthesis that would be prescribed for a person of similar height and weight.

DETAILED DESCRIPTION:
Subject Selection and Consent:

Subjects will be selected based on the following priority. Subjects who have previously participated in similar studies with the Biomechatronics lab and who have already been screened for health and mobility level will be contacted first. If additional subjects are needed, a recruitment flyer and screening questionnaire will be sent to potential candidates. Copies of both the flyer and questionnaire are included in the attachments section. Prior to the experimental sessions, subjects will be asked to read and sign a informed consent form and will explain the project to them and answer any questions that they may have. They will also be given time to become familiar with the equipment being used before beginning any trials. If needed, subjects will be aligned and fitted by a professional prosthetist at A Step Ahead Prosthetics in Burlington, MA. No personnel at A Step Ahead Prosthetics will conduct research or have any vested interest in research outcomes or publication.

Attire:

Subjects will be asked to wear tight-fitting clothes, such as a skin-tight shirt, running shorts and low-profile shoes. If this is not possible, clothes will be provided according to subject needs. The investigators will provide and may require subjects to wear a skin-tight Velcro outfit that allows us to place reflective balls for video camera capture.

Location(s) and Timeline:

Experimental sessions will be conducted in the MIT Biomechatronics Laboratory (E14-274), 75 Amherst St., Cambridge, MA 02139. Any alignment and fitting of prosthetic devices will take place at A Step Ahead Prosthetics, 21 A. St., Burlington, MA 01803.

Total study duration is expected to be 8 hours per subject, likely over two 4-hour sessions. These sessions can be completed either in a single day or over two days. After subject selection, the entire study is expected to take 3 months.

Powered Prosthesis:

Subjects will be given two computer-controlled, powered ankle-foot prostheses to attach in place of their customary prosthesis during a session. These include the Blatchford Elan as well as a variable-stiffness prosthesis developed in the Biomechatronics lab. These powered prostheses have the capability of providing active assistance or changing mechanical properties during walking. Controls can be adjusted either through a wireless link or hardwire connection depending on the device. Subjects will be given as much time as necessary to practice using the prostheses before the experiments begin.

Passive Prosthesis:

Subjects will be given three passive prostheses to attach in place of your customary prosthesis during a session. These include the Ossur Pro-flex XC, a passive sliding-beam prosthesis, and a passive prosthesis that can change ankle equilibrium angle manually. Subjects will be given as much time as necessary to practice using the prosthesis before the experiments begin.

Data Collection:

Data collection is expected to take place in two segments. The first segment consists of level-ground walking on a treadmill at three speeds between 0.5-1.5m/s (slow to fast walking). At each speed, all five prostheses will be tested, randomly selected, for 2mins each. Motion will be captured with a VICON motion capture system, and ground reaction forces will be measured using a Bertec force-sensitive treadmill. For each speed, once all prostheses have been tested, each subject will be given a questionnaire to ascertain how each prosthesis performed at heel strike (early stance), roll over (mid stance), and powered plantar flexion (late stance). In addition, each subject will be asked how each prosthesis generally performed, and their personal preference. This testing will occur across the three walking speeds, resulting in three completed questionnaires.

In addition, subjects will walk in a figure-8 pattern at a preferred gait speed around two cones placed on the level-ground walking surface and separated by up to 30 feet. Subjects will perform the walking figure-8 for a minimum of 5 times for each randomly-selected prosthesis. Once all prostheses have been tested, each subject will be given a questionnaire to ascertain how each prosthesis generally performed, and their personal preference.

The second session will consist of slope and stair walking. Each subject will ascend and descend stairs and a ramp inclined between 4°-10° from horizontal at their preferred speed, in a randomly selected order. Motion will be captured with a VICON motion capture system, and ground reaction forces will be measured using a Bertec force-sensitive treadmill for slope ambulation, and a force-sensitive staircase for stair ambulation. All five prostheses will be tested, randomly selected. Subjects will perform each of stair ascent and stair descent for a minimum of 5 times per prosthesis. For slope ambulation on an instrumented treadmill, subjects will walk for a total of 2mins for slope ascent and 2mins for slope descent with each prosthesis. For each slope and stair ascent/descent, once all prostheses have been tested, each subject will be given a questionnaire to ascertain how each prosthesis generally performed, and their personal preference. This testing will occur across the slope terrain types, as well as after the stair ascent/descent trial, resulting in three completed questionnaires for each subject.

ELIGIBILITY:
Inclusion Criteria:

* Person with unilateral transtibial amputation
* K3 or K4 Medicare mobility rating
* Ages 18-65

Exclusion Criteria:

* Below K3 Medicare mobility rating
* Outside of age range (liability and safety reasons)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
User device preference for level-ground walking | From enrollment to the end of trial (2 sessions, 8 hours total per patient)
  Determine which device the users prefer for level-ground walking by gauging user feedback through an evaluation questionnaire. Evaluation units will be a sliding scale ranging from "Very unfavorable" to "Very favorable" with neutral in the middle. Subjects will be asked to rank the 5 interventions from best to worst for the specific task.
User device preference for stair ascent & descent | From enrollment to the end of trial (2 sessions, 8 hours total per patient)
  Determine which device the users prefer for stair ascent & descent by gauging user feedback through an evaluation questionnaire. Evaluation units will be a sliding scale ranging from "Very unfavorable" to "Very favorable" with neutral in the middle. Subjects will be asked to rank the 5 interventions from best to worst for the specific task.
User device preference for sloped ground ascent & descent | From enrollment to the end of trial (2 sessions, 8 hours total per patient)
  Determine which device the users prefer for 8-degree sloped ground ascent & descent by gauging user feedback through an evaluation questionnaire. Evaluation units will be a sliding scale ranging from "Very unfavorable" to "Very favorable" with neutral in the middle. Subjects will be asked to rank the 5 interventions from best to worst for the specific task.

SECONDARY OUTCOMES:
Effect of device on level-ground walking gait | From enrollment to the end of trial (2 sessions, 8 hours total per patient)
  Evaluate the effect of the device on level-ground walking gait patterns. Gait will be measured with a VICON motion capture system. Unit of measure is gait symmetry.
Effect of device on stair ascent & descent gait | From enrollment to the end of trial (2 sessions, 8 hours total per patient)
  Evaluate the effect of the device on stair ascent and descent gait patterns. Gait will be measured with a VICON motion capture system. Unit of measure is gait symmetry.
Effect of device on sloped ground walking gait | From enrollment to the end of trial (2 sessions, 8 hours total per patient)
  Evaluate the effect of the device on sloped ground walking gait patterns. Gait will be measured with a VICON motion capture system. Unit of measure is gait symmetry.
Effect of device on ground reaction force during ambulation | From enrollment to the end of trial (2 sessions, 8 hours total per patient)
  Evaluate the effect of the device on ground reaction forces during ambulation. Ground reaction forces will be measured with Bertec force plates. Unit of measure is ground reaction force in Newtons.

CONTACTS AND LOCATIONS:
Locations (1):
- MIT Media Laboratory, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/55/NCT05964855/ICF_000.pdf